CLINICAL TRIAL: NCT06593652
Title: Evaluating Caregiver Involvement in Primary Care-Based Brief Interventions for Adolescent Alcohol Use Problems
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Principal Investigator, Zachary W. Adams, Associate Professor, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23394
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-10

CONDITIONS: Alcohol Use; Adolescent; Mild Alcohol Use Disorder; Mild Substance Use Disorder
Keywords: Brief Intervention; Teen Intervene; Caregiver Involvement; Alcohol Use; Substance Use
MeSH Terms: conditions — Alcohol Drinking; Substance-Related Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The data analysts will be masked to intervention condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Teen Intervene - Adolescent Only (Active Comparator): Only the youth will participate in the brief intervention, Teen Intervene. The youth will participate in manual-standardized Teen Intervene sessions.
  Interventions: Behavioral: Teen Intervene - Adolescent Only
- Teen Intervene - Caregiver Involvement (Experimental): The youth will participate in two Teen Intervene sessions. Additionally, the caregiver(s) will participate in a single, caregiver-only Teen Intervene session.
  Interventions: Behavioral: Teen Intervene with Caregiver Session
- Teen Intervene - Online Caregiver Support Tool (Experimental): Only the youth will participate in the brief intervention, Teen Intervene. The youth will participate in two Teen Intervene sessions. Caregiver(s) will be provided with an online tool (Family Checkup Online) that addresses parenting strategies to support their youth.
  Interventions: Behavioral: Family Check Up

INTERVENTIONS:
Behavioral: Teen Intervene - Adolescent Only — Teen Intervene (TI) is delivered over two or three, 45- to 60-minute sessions (2 teen sessions +/- 1 caregiver session) to reduce youth substance use, increase motivation for abstinence, and promote use of existing coping strategies. TI is an adolescent-appropriate adaptation of motivational enhancement therapy (MET), and includes a discussion of readiness to change, goal setting, personal feedback, a functional analysis of substance use, and a review of coping skills.
  Arms: Teen Intervene - Adolescent Only
Behavioral: Teen Intervene with Caregiver Session — Teen Intervene (TI) is delivered over two or three, 45- to 60-minute sessions (2 teen sessions +/- 1 caregiver session) to reduce youth substance use, increase motivation for abstinence, and promote use of existing coping strategies. TI is an adolescent-appropriate adaptation of motivational enhancement therapy (MET), and includes a discussion of readiness to change, goal setting, personal feedback, a functional analysis of substance use, and a review of coping skills. In this condition, the caregiver session will address caregiver expectations around youth substance use and strategies for promoting positive youth behavior change including reduced substance use.
  Arms: Teen Intervene - Caregiver Involvement
Behavioral: Family Check Up — Family Check-Up Online (FCU-O) is a self-paced, parent-driven, fully HIPAA compliant online version of the Family Check-Up (FCU), a brief intervention that integrates assessment, motivation-enhancement, and skill building to help parents effectively manage behavior and build positive relationships with their children aged 2-17 in order to reduce emotional and behavioral problems among youth.
  Arms: Teen Intervene - Online Caregiver Support Tool

SUMMARY:
Intervention for mild severity alcohol use among U.S. teens is crucial, as alcohol is the most commonly used substance in this age group, yet few receive the necessary interventions. Primary care, where over 90% of youth regularly visit, is an ideal setting for identifying and addressing mild alcohol use disorder (AUD) through brief interventions like motivational interviewing (MI) and cognitive-behavioral therapy (CBT). However, for teens with mild AUD, a single brief session may not be sufficient, raising questions about the role of caregiver involvement. This study seeks to determine the most effective level of caregiver involvement-no involvement, a single live session, or an online self-paced program-in reducing alcohol use among adolescents with mild AUD in primary care settings. The study also explores the impact of these interventions on other outcomes such as substance use and psychosocial functioning, as well as the factors influencing treatment response. The results will guide the selection and implementation of effective, scalable interventions in primary care to address youth alcohol use disorders.

DETAILED DESCRIPTION:
Detailed Description

Intervention for mild severity alcohol use is needed in primary care. Alcohol is the most commonly used substance among U.S. teens (lifetime use: 62% of 12th graders) and contributes to myriad harms, yet few youth who may benefit from intervention ever receive it. Primary care is an ideal setting for identifying and delivering brief interventions to youth with mild severity alcohol problems since over 90% of youth attend primary care visits routinely and substance use screening is standard practice. For youth with infrequent, low-risk use, brief (15-30 minute) motivational conversations may be sufficient to reduce risk. In contrast, youth with moderate to severe alcohol problems typically require more intensive interventions delivered by behavioral health specialists (e.g., intensive outpatient, residential treatment). A critical decision faced in primary care settings is what to do for youth who fall between these ends of the spectrum-namely, youth who show early signs of problematic use, meeting criteria for mild severity alcohol use disorder (AUD) (i.e., 2-3 symptoms; estimated to be approximately 3% of youth aged 12-17). Strong evidence supports individual-level brief interventions that incorporate motivational interviewing (MI) and basic cognitive-behavioral therapy (CBT) skills to help youth reduce substance use frequency, volume, and related impairment among youth with mild AUD.

Caregiver involvement in brief interventions for mild severity AUD may improve outcomes. Systematic reviews support interventions that address family-level factors (e.g., parents' attitudes, parenting behavior). When and how to involve parents or other primary caregivers in interventions for youth with mild severity AUD remains unclear. For instance, in a large school-based trial, brief MI+CBT without a caregiver session was equivalent to brief MI+CBT with a caregiver session on alcohol outcomes and drug consequences, whereas the MI+CBT with a caregiver session modestly outperformed the adolescent-only condition on cannabis-related outcomes.

Directly intervening with caregivers can be difficult and impractical. Despite the potential benefits of caregiver involvement, many caregivers see their child's behavior and choices as the main concern and therefore may be less inclined to participate in services focused exclusively on parenting practices. Caregivers may also have to miss work for parenting-dedicated sessions, which can disproportionately impact economically disadvantaged families. Asynchronous online programming may address some of these barriers-and preliminary findings support acceptability and efficacy of this approach-but such programs remain understudied relative to more traditional program structures. Identifying the relative effectiveness of online versus in-person caregiver components compared to youth-only interventions is critical to support decisions and eventual cost-benefit analyses about which programs to offer to different patients.

The primary research question this study aims to address is, "What type and level of caregiver involvement in a brief youth-focused intervention (i.e., Teen Intervene) results in the greatest reductions in alcohol use among adolescents with mild alcohol use disorder when delivered in a primary care context: no caregiver involvement, a single dedicated parent session, or a self-paced online parenting program?" Secondary research questions are "What is the relative impact of the three intervention models on other substance, academic, and behavioral health outcomes?" and "Do youth (i.e., personality, alcohol/substance risk perceptions, etc.) and family factors (i.e., parental monitoring) moderate treatment response?" Understanding implementation factors associated with each intervention is also of interest, as engaging caregivers in youth SUD services can be challenging. Thus, the outcomes of the current project will help inform the selection and delivery of interventions that are both effective and reasonable to implement in primary care contexts, where most youth receive healthcare services. When delivered at scale, such interventions could help address the alcohol and other substance use disorders affecting the U.S. today.

Specific Aims

A Type 1 hybrid effectiveness-implementation trial is proposed to compare the effectiveness of an individual skill-building MI+CBT brief intervention (Teen Intervene, TI) with varying caregiver involvement: a) no caregiver involvement, b) a single live caregiver session, and c) an online, self-paced parenting program (Family Check-Up Online, FCU). These brief intervention programs will be tested as a first-level intervention to address mild AUD and prevent progression to more severe AUD symptoms or patterns of use. The aims are two-fold:

Aim 1: Compare the effectiveness of a youth-focused brief intervention (TI) when delivered without caregiver involvement (TI-A) versus with an added caregiver session (TI-A+P) versus with an online caregiver component (TI-A+FCU) in reducing alcohol use in adolescents with mild AUD in primary care. The overall magnitude of response and percentage of youth in each condition with clinically meaningful changes (i.e., % responders) will be measured. It is predicted that TI-A+P > TI-A+FCU > TI-A. Secondary outcomes will include other substance use (e.g., vaping, cannabis), AUD/SUD symptoms, general psychosocial functioning, and implementation factors including reactions to the intervention (e.g., satisfaction, acceptability, barriers).

Aim 2: Identify youth and family factors associated with intervention response versus non-response in each treatment condition, such as baseline substance use intensity (frequency, volume, duration, type), youth and caregiver perception of alcohol/substance use risk, youth personality factors (impulsivity, emotion dysregulation), and baseline parenting practices. Intervention implementation factors will also be examined. This aim will be accomplished through both quantitative and qualitative measures.

ELIGIBILITY:
Inclusion Criteria:

* 12-17 years old;
* Mild to moderate severity for alcohol use (based on standardized surveys from their primary care provider or clinical indication) or other substance use
* English language fluency

Exclusion Criteria:

* N/A

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 615 (Estimated)
Dates: Start 2025-08-19 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Timeline Follow-Back | *0-at time of intervention, *3 months after time of intervention; *6 months after time of intervention; *12 months after time of intervention
  30 items that assess daily alcohol usage over the past month will be administered to all participants. Participants will be queried about number of standard drinks consumed each day.

SECONDARY OUTCOMES:
Timeline Follow-Back | *0-at time of intervention, *3 months after time of intervention; *6 months after time of intervention; *12 months after time of intervention
  30 items that assess other substance usage over the past month will be administered to all participants. Participants will be queried about amount of each substance used for each day.
DAST-A | *0-at time of intervention, *3 months after time of intervention; *6 months after time of intervention; *12 months after time of intervention
  28 items that review AUD/SUD symptoms will be administered to all participants.
SUD Services Engagement | *0-at time of intervention, *3 months after time of intervention; *6 months after time of intervention; *12 months after time of intervention
  14 items that review youths services received by the participant (e.g., mental health treatment, substance use treatment, hospitalization) over the past 3 months per caregiver report. This will be asked to all participant caregivers.
PROMIS Surveys | *0-at time of intervention, *3 months after time of intervention; *6 months after time of intervention; *12 months after time of intervention
  37 items that review Psychosocial Functioning (Peer Relationships, Life Satisfaction, Depression, Anxiety, Anger/Irritability, and Psychological Stress Experiences). These items will be administered to all participants.

OTHER OUTCOMES:
Client Satisfaction Questionnaire | *0-at time of intervention, *3 months after time of intervention; *6 months after time of intervention; *12 months after time of intervention
  8 items that assesses adolescent/caregiver-reported implementation factors
Communities That Care Survey Family Factors | *0-at time of intervention, *3 months after time of intervention; *6 months after time of intervention; *12 months after time of intervention
  38 items that assesses family/caregiver practices
Acceptability, Feasibility, and Appropriateness of Intervention Measure | once a year
  8 items that assesses interventionist-reported implementation factors

CONTACTS AND LOCATIONS:
Overall Officials: Zachary Adams, PhD, HSPP, Principal Investigator — Indiana University; Tamika Zapolski, PhD, HSPP, Principal Investigator — Indiana University
Locations (1):
- IU Health/Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Though the researchers are not required to provide information about plans to share individual participant data (IPD), we plan to withhold individual participant data from sharing. This decision aligns with university policy and the terms outlined in our participants' consent forms, which stipulate that patient information will not be shared publicly.